CLINICAL TRIAL: NCT04882033
Title: An Exploratory Clinical Study to Investigate Concurrent Chemoradiotherapy Combination With Anlotinib for Limited-stage Small Cell Lung Cancer
Brief Title: Concurrent Chemoradiotherapy Combination With Anlotinib for Limited-stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L039
Record Dates: First submitted 2021-05-07; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2020-05

CONDITIONS: Small Cell Lung Cancer Limited Stage
MeSH Terms: interventions — Chemoradiotherapy; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent chemoradiotherapy plus anlotinib (Experimental): Concurrent chemoradiotherapy plus anlotinib for 4-6 cycles This study will include a sequential evaluation of 3 subjects per dose group. Low-dose groups: anlotinib 8mg per day with concurrent chemoradiotherapy. Middle-dose groups: anlotinib 10mg per day with concurrent chemoradiotherapy. High-dose groups: anlotinib 12mg per day with concurrent chemoradiotherapy.
  Interventions: Drug: Concurrent chemoradiotherapy plus anlotinib

INTERVENTIONS:
Drug: Concurrent chemoradiotherapy plus anlotinib — Anlotinib: for cycle 1-6. P.O; QD; from days 1 to 14 in a 21-day cycle. 8mg in low-dose groups (3 subjects). 10mg in middle-dose groups (3 subjects). 12mg in high-dose groups (3 subjects).
  Chemotherapy:
  For cycle 1/4/5/6. Etoposide 100mg/m2, d1-3, q3w; Cisplatin 25mg/m2 d1-3, q3w. For cycle 2/3. Etoposide 50mg/m2, d1-3, q4w; Cisplatin 25mg/m2 d1-3, q4w.
  Radiotherapy:
  For cycle 2/3.Thoracic radiotherapy dose will be 2.0Gy per day, given 5 days a week, to cumulative dose of 60～66Gy.

SUMMARY:
The purpose of this study is to evaluate the tolerability and toxicity of different dose of anlotinib combination with concurrent chemoradiotherapy in the treatment of limited-stage SCLC patients.

DETAILED DESCRIPTION:
Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR1、VEGFR2、VEGFR3、FGFR1/2/3、PDGFRa/β c-Kit and MET. The purpose of this study is to determine the maximum tolerated dose of anlotinib when combination with concurrent chemoradiotherapy. From low dose group up to high dose group, each one had 3 patients at least. Primary group received anlotinib 8mg. The dose of anlotinib would increase gradually until MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, signed informed consent.
2. Patients aged between 18 -75 years; According to the eighth edition of AJCC and the standard of the VALG two-stage staging method, the patient is confirmed by histology or cytology as limited-stage SCLC (stage I-III, any T, any N, M0) and cannot be operated on.
3. Patients with ECOG PS Scoring: 0~1 point
4. Patients with concurrent chemoradiotherapy must comply with relevant regulations.
5. PCI is given according to the judgment of the investigator.
6. Patients with normal organ function, the following criteria are met: (1) blood routine examination criteria (without blood transfusion in 14 days) : a) hemoglobin (HB) ≥90g/L; b) absolute neutrophil count (ANC) ≥1.5×10e9/L; c) platelet (PLT) ≥80×10e9/L; (2) biochemical tests meet the following criteria: a) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); b) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN, if liver metastasis occurred, ALT and AST ≤5 ULN; c) serum creatinine (Cr) ≤1.5 ULN or creatinine clearance (CCr) ≥60mL/min.
7. For women of child-bearing age, the pregnancy test results (serum or urine) within 1 week before enrolment must be negative. They will take appropriate methods for contraception during the study until the 6 months post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 6 months post the last administration of study drug.

Exclusion Criteria:

1. Small cell and non-small cell mixed lung cancer
2. Extensive stage small cell lung cancer
3. Central lung tumors that imaging shows tumor lesions invade local large blood vessels; or with significant pulmonary cavum or necrotizing
4. Less than 4 weeks from the last clinical trial or participating in other clinical studies.
5. History:

1) Brain metastasis or spinal cord compression 2) Other active malignancies that require simultaneous treatment. 3) History of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or history of organ transplantation.

4) History of mental drug abuse and cannot be cured or have mental disorders 6. Patients with any severe and/or uncontrolled disease, including:

1. blood pressure control is not ideal (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg);
2. Significant cardiac disease as defined as: grade I or greater myocardial infarction, unstable arrhythmia (including corrected QT interval (QTc ) period between male or greater 450 ms, female or greater 470 ms); New York Heart Association (NYHA) grade II or greater heart dysfunction , or Echocardiography reveal left ventricular ejection fraction (LVEF) less than 50%
3. Decompensated diabetes or other remedies for high-dose glucocorticoid therapy.
4. Exacerbation of chronic obstructive pulmonary disease (COPD) or other serious respiratory diseases that require hospitalization
5. Active or uncontrollable serious infection (≥CTC AE Level 2 infection);
6. Uncontrolled pleural effusion, pericardial effusion and abdominal effusion requiring repeated drainage.
7. Urine routine test protein≥++, and confirmed 24 hours urine protein>1.0 g; 7. Imaging shows that the tumor has been violated around important vascular or the researchers determine the tumor is likely to invade important blood vessels caused by fatal bleeding during the follow-up.

8. Patients who received a major surgical treatment or severe trauma, the effects of surgery or trauma have been eliminated in less than 2 weeks before being enrolled 9. Patients with clinically significant hemoptysis occurred within 3 months prior to enrollment (greater than 1/2 teaspoon of bright red blood). History of clinically relevant major bleeding event (e.g. gastrointestinal hemorrhage, hemorrhagic acne, bleeding gastric ulcer, occult blood test ≥ ++, or vasculitis, etc.) 10. Patients who have arterial/venous thromboembolism events within 6 months before being enrolled, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.

11. Coagulation disfunction（INR>1.5 or PT>upper limit of normal(ULN)+4s or activated partial thromboplastin time (APTT) >1.5 upper limit of normal (ULN)）, hemorrhagic tendency or receiving the therapy of thrombolysis or anticoagulation.

12. At the discretion of the investigator, the patient may have other factors that may cause the study to be terminated midway.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-05-07 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerance Dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DLT reported. | From enrollment to completion of study. Estimated about 18months
  Dose Limiting Toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.03 criteria

SECONDARY OUTCOMES:
PFS（Progress free survival） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  The PFS time is defined as time from enrollment to locoregional or systemic
OS（Overall Survival） | From enrollment until death (up to 24 months)
  OS was defined as time from date of enrollment to date of death due to any cause.
ORR（Objective Response Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.
DCR（Disease Control Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individal participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requesdtors will be required to sign a Data Access Agreement.
URL: http://www.cttq.com/